CLINICAL TRIAL: NCT04521036
Title: Assessment of the Safety and Efficacy of Convalescent Plasma to Treat COVID-19 Patients With Moderate and Above Illness
Brief Title: Convalescent Plasma for COVID-19 Patients (CPCP)
Acronym: CPCP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other); National Hospital for Tropical Diseases, Hanoi, Vietnam (Other Government); National Institute of Hematology and Blood Transfusion, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISC.20.11.2
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: COVID 19
MeSH Terms: conditions — COVID-19 | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This trial is a randomized comparative trial. Patients will be randomized between the infusion of 500mL of Convalescent Plasma versus the standard of care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convalescent plasma (Experimental): Standard of care plus 500 mL of convalescent plasma from COVID-19 recovered donors
  Interventions: Biological: Convalescent Plasma as Therapy for Covid-19 patients
- Standard of care (No Intervention): Standard of care (Supportive care, oxygen, antibiotics, no convalescent plasma)

INTERVENTIONS:
Biological: Convalescent Plasma as Therapy for Covid-19 patients — Patients in the treatment group will receive 500 ml from COVID-19 recovered donors
  Arms: Convalescent plasma

SUMMARY:
Prior findings in various viral respiratory diseases including SARS-CoV-related pneumonia suggest that convalescent plasma can reduce mortality, although formal proof of efficacy is still lacking. The investigators propose to evaluate intravenous administration of convalescent plasma (CP) obtained from COVID19 survivors in COVID19 patients who are in the medium stage. Supportive data exist for use of convalescent plasma in the treatment of COVID19 and other overwhelming viral illnesses. The study team wants to test the hypothesis that treatment with COVID19 CP will demonstrate salutary effects on COVID19 disease severity/duration, with the primary objective to reduce mortality. In addition, a major secondary objective to reduce the requirement for and/or duration of mechanical ventilation. This phase is to test the safety and efficacy of CP therapy.

DETAILED DESCRIPTION:
Coronaviruses are among the most common causes of the common cold in humans. In recent decades, coronavirus has caused several epidemics worldwide with a vast number of deaths such as severe acute respiratory syndrome-SARS (2003) with 8098 people infected, and 774 people died over 29 countries. The disease caused by SARS CoV-2 (COVID19) is manifest by fever, fatigue, dry cough, pharyngitis, and headache. In addition to the common clinical presentation of respiratory distress, and increasing frequency of cardiovascular manifestations has become evident.

In this context, the investigators propose to evaluate the safety and efficacy of intravenous administration of convalescent plasma (CP) obtained from COVID19 survivors in patients requiring hospitalization for symptomatic "high risk" COVID19 disease. The study team wants to test the hypothesis that treatment with COVID19 CP will demonstrate salutary effects on COVID19 disease severity/duration, with the primary objective to reduce mortality. In addition, a major secondary objective to reduce the requirement for and/or duration of mechanical ventilation. This is a randomized clinical trial comparing convalescent plasma with the standard of care therapy in patients hospitalized for COVID-19 in Vietnam. Patients were randomized 1:1 and received 500 ml of plasma with anti-SARSCoV-2 neutralizing antibody titers of at least 1:80.

Written informed consent will be obtained all eligible subjects prior to participation.

Convalescent plasma will be obtained from male donors, nulliparous females, or female donors negative for HLA antibodies at least 14 days following recovery from COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* SARS-CoV-19 PCR positive
* Moderate stage and above
* Time from onset to screening ≤ 21 days, the SARS-CoV-2 test is still positive

Exclusion Criteria:

* Patients with a history of autoimmune disease or IgA deficiency
* Patients with a history of allergy
* Multi-organ/system failure
* Pregnant or breastfeeding at the time of study
* Cancer, history of heart failure, stroke, bronchial asthma
* Multi-organ/system failure with indications for dialysis, severe hypoxia, failure with conventional treatment methods, indications for ECMO.
* The patient is infected with multidrug-resistant bacteria.
* The patient is participating in another study.
* Time from onset to screening> 21 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Change in mortality | until hospital discharge or a maximum of 60 days whichever comes first
  Change in mortality of high risk COVID 19 disease compared with the control arm

SECONDARY OUTCOMES:
Change in requirement for mechanical ventilation | until hospital discharge or a maximum of 60 days whichever comes first
  Change in the duration of mechanical ventilation in high risk COVID 19 disease compared with the control arm
Change in the duration of mechanical ventilation | until hospital discharge or a maximum of 60 days whichever comes first
  Change in the time a participant will remain on the ventilator
Incidence of Treatment-Emergent Adverse Events | Incidence of Treatment-Emergent Adverse Events until hospital discharge or a maximum of 60 days whichever comes first
  Incidence of Treatment-Emergent Adverse Events during study period

CONTACTS AND LOCATIONS:
Overall Officials: Liem Thanh Nguyen, PhD, Principal Investigator — Vinmec Research Institute of Stem Cell and Gene Technology
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No